CLINICAL TRIAL: NCT07106047
Title: Empowering Asthmatic Seniors: Nursing Interventions to Mitigate Climate Change-related Effects on Symptom Severity and Physical Capacity
Brief Title: Nursing Interventions to Mitigate Climate Change-related Effects on Asthma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norther Private Collage of Nursing (Other)
Collaborators: Minia University (Other)
Responsible Party: Principal Investigator, Amal Hashem, Associate professor, Norther Private Collage of Nursing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Asthmatic senior
Record Dates: First submitted 2025-07-25; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Elsner's Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nurse-Led Climate-Responsive Asthma Management Program (Experimental): Participants in this arm will receive a structured, nurse-led intervention designed to reduce asthma symptom severity and maintain physical capacity in older adults during climate change-related environmental stressors such as extreme heat or poor air quality.
  The intervention includes:
  Personalized Asthma Action Plan tailored to the individual's triggers and medication regimen.
  Environmental Exposure Education on recognizing and responding to climate-related asthma triggers (e.g., heat, pollen, pollution).
  Weekly Nurse Coaching Sessions (30-45 minutes via phone or in-person) for 12 weeks, focusing on self-management strategies, symptom tracking, inhaler technique, and physical activity guidance.
  Distribution of Support Tools, including peak flow meters, symptom diaries, and access to real-time air quality alerts.
  Physical Activity Modification Plans developed with nursing staff to maintain mobility while minimizing risk during high-pollution or extreme weather days.
  Interventions: Behavioral: Nurse-Led Climate-Responsive Asthma Management Program

INTERVENTIONS:
Behavioral: Nurse-Led Climate-Responsive Asthma Management Program — A structured behavioral intervention delivered by trained nurses, focusing on climate-adapted asthma self-management for older adults. The program includes personalized coaching on symptom monitoring, environmental risk response, inhaler technique, and safe physical activity planning during climate stress events. Intervention is delivered weekly over 12 weeks through a combination of phone and in-person sessions, supported by tools such as symptom diaries, air quality alerts, and peak flow meters.
  Other Names: Climate-Smart Asthma Care for Seniors

SUMMARY:
This study aims to evaluate the effectiveness of targeted nursing interventions in reducing asthma symptom severity and improving physical capacity among older adults during periods of heightened environmental stress caused by climate change (e.g., heat waves, poor air quality). By equipping seniors with practical self-management strategies and personalized support, the study seeks to enhance resilience against climate-related health risks and promote overall well-being.

DETAILED DESCRIPTION:
Climate change has increasingly been linked to the worsening of chronic respiratory conditions, particularly among vulnerable populations such as older adults with asthma. Rising temperatures, extreme weather events, and elevated air pollution levels pose serious health threats by exacerbating symptoms and limiting physical activity.

This interventional study focuses on developing and implementing a nursing-led, community-based support model that empowers asthmatic seniors to better manage their condition amid climate change stressors. The intervention includes personalized asthma action plans, environmental exposure education, physical activity guidance, and symptom monitoring tools. Participants will receive individualized coaching from trained nurses to build adaptive behaviors that reduce symptom severity and maintain physical capacity during adverse environmental conditions.

Primary outcomes include changes in asthma symptom scores, physical function (e.g., six-minute walk test), and quality of life metrics. Secondary outcomes include frequency of asthma exacerbations, healthcare utilization, and adherence to preventive behaviors.

The study underscores the role of nursing in advancing climate-resilient care models that address the health needs of aging populations in an increasingly volatile environment.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 65 years and older

Clinically diagnosed with asthma (physician-confirmed)

Stable asthma (no hospitalizations for asthma in the past 30 days)

Able to understand and provide informed consent

Willing and able to participate in a 12-week nursing intervention program

Has access to a telephone or internet-enabled device for coaching sessions and monitoring

Resides in an area prone to climate-related environmental stressors (e.g., urban heat, poor air quality)

Exclusion Criteria:

Diagnosis of chronic obstructive pulmonary disease (COPD) or other significant pulmonary conditions (e.g., interstitial lung disease)

Severe cognitive impairment (e.g., diagnosed dementia) that would interfere with participation

Current participation in another asthma-related interventional study

Residing in long-term care facilities where independent asthma self-management is not feasible

Any unstable medical condition that could confound outcomes or pose safety risks, as determined by the study physician

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in Asthma Symptom Severity Score | Baseline and 12 weeks post-intervention
  Assessed using a validated instrument such as the Asthma Control Test (ACT), this outcome measures the change in asthma symptom severity from baseline to the end of the intervention period. A higher ACT score indicates better asthma control.